CLINICAL TRIAL: NCT01146626
Title: Does Vitamin D Supplement Improve SVR in Chronic Hepatitis C (Genotype 2,3) in naïve Patients Treated With Peginterferon Alpha and Ribavirin
Brief Title: Does Vitamin D Improves Sustained Virologic Response (SVR) in Genotype 2,3 Chronic Hepatitis C Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Collaborators: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Liver Clinic, Ziv medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV +Vitamin D
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2010-06

CONDITIONS: Hepatitis C
Keywords: Vitamin D; Hepatitis C; Genotype2,3; SVR; Naive; RVR rate; EVR rate; SVR rate
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peg+ Vitamin D+ Ribavirine (Active Comparator): Peg+ Vitamin D+ Ribavirine
  Interventions: Drug: Peg+ Vitamin D+ Ribavirine
- Peg+ Ribavirine (Experimental): Peg+ Ribavirine
  Interventions: Drug: Peg+ Ribavirine

INTERVENTIONS:
Drug: Peg+ Vitamin D+ Ribavirine — Peg+ Vitamin D+ Ribavirine
  Arms: Peg+ Vitamin D+ Ribavirine
Drug: Peg+ Ribavirine — Peg+ Ribavirine
  Arms: Peg+ Ribavirine

SUMMARY:
Standard therapy for chronic hepatitis C virus (HCV) is (Peg/RBV) combination therapy obtaining sustained virologic response (SVR) in 80% of naïve patients with genotype 2,3. Studies rarely address the issues of improving host factors. The current study examines

1. whether adding vitamin D, a potent immunomodulator, could improve viral response and shorten treatment duration (from 24 weeks to 12 weeks)
2. whether Vitamin D levels predictes negative treatment outcome.

DETAILED DESCRIPTION:
Standard therapy for chronic hepatitis C virus (HCV) is (Peg/RBV) combination therapy obtaining sustained virologic response (SVR) in 80% of naïve patients with genotype 2,3. Studies rarely address the issues of improving host factors. The current study examines whether adding vitamin D, a potent immunomodulator, could improve viral respons.The working hypothesis is that Adding vitamin D to conventional Peg/RBV therapy for naïve, genotype 2,3 patients with chronic HCV infection significantly improves RVR, EVR, and SVR

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age,
* Chronic genotype 2,3 HCV infection, Traetment Naive
* Negative sero for HBV, HDV and HIV viral infections
* Absolute neutrophil count of >1500 per cubic millimeter, a platelet count of >90,000 per cubic millimeter
* Normal hemoglobin level

Exclusion Criteria:

* Decompensated liver disease (cirrhosis with CP score >9)
* Another cause of clinically significant liver disease
* Hepato cellular carcinoma
* Psychiatric Disorder
* Chronic heart failure
* Pregnant women
* Uncontrolled diabetes with retinopathy
* Arythmia
* Active CAD
* Positive sero for HBV, HDV and HIV viral infections or other autoimmune liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-02 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
SVR rate | 1 year
  to evaluate the response rate

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Liver clinic, Hedera
  - Ziv medical center liver unit, Safed, Israel